CLINICAL TRIAL: NCT00293241
Title: PreFER MVP for Elective Replacement
Brief Title: PreFER Managed Ventricular Pacing (MVP) For Elective Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 2-Aug 21, 2007
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Cardiovascular Diseases
Keywords: Pacemaker or ICD replacement
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MVP ON (Other): Managed Ventricular Pacing programmed on
  Interventions: Device: Managed Ventricular Pacing programmed ON/OFF
- MVP OFF (Other): Managed Ventricular Pacing programmed off: conventional pacing
  Interventions: Device: Managed Ventricular Pacing programmed ON/OFF

INTERVENTIONS:
Device: Managed Ventricular Pacing programmed ON/OFF — Device programming

SUMMARY:
The purpose of this study is to demonstrate the benefit of MVP in pacemaker and implantable cardioverter defibrillator (ICD) patients with a history of right ventricular pacing.

DETAILED DESCRIPTION:
A number of clinical studies (Danish I, Danish II, David, MOST) over the past few years have shown that, in patients with intact atrioventricular (AV) conduction, unnecessary chronic right ventricular (RV) pacing can cause a variety of detrimental effects, including atrial fibrillation (AF), left ventricular (LV) dysfunction, and congestive heart failure (CHF). These effects are believed to result from the mechanical dyssynchrony and ventricular chamber dysfunction that occurs with chronic, single-site, apical ventricular stimulation.

Therefore a new pacing modality, Managed Ventricular Pacing (MVP), was designed to give preference to natural heart activity by minimizing unnecessary right ventricular pacing. This is accomplished by automatically switching between single chamber atrial and dual-chamber pacing based on specific patient needs.

MVP is an atrial-based dual-chamber pacing mode that provides functional AAI/R pacing with ventricular monitoring and back-up DDD/R pacing only as needed during episodes of AV block.

The reversibility of the detrimental effects caused by ventricular pacing has been initially investigated in small patient populations with short pacing durations in AAI and needs further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a dual chamber device (including atrial synchronous ventricular inhibited [VDD]) for a minimum time duration of 2 years
* Planned to be replaced or replaced with a device including the MVP feature
* Have had more than 40% ventricular pacing documented with their old device over a period of at least 4 weeks before enrollment or device replacement.
* Pacing should not be caused by a switch to the single chamber pacing (VVI) mode because of battery depletion
* Have signed the informed consent
* Have no need to change the pacing mode or the atrioventricular (AV) intervals.

Exclusion Criteria:

* Patients with a cardiac resynchronization therapy (CRT) indication
* Permanent AF
* Permanent AV block
* Inability to complete follow-up visits at a study center.
* Unwillingness or inability to cooperate or give written informed consent, or the patient is a minor, and legal guardian refuses to give informed consent
* Planned cardiovascular intervention
* Inclusion in another clinical trial that will affect the objectives of this study
* Neurocardiogenic syncope as primary implantable pulse generator (IPG) indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2006-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Piot, Dr., Principal Investigator — Centre Cardiologique du Nord, Saint-Denis, France; Aurelio Quesada, Dr., Principal Investigator — Hospital General Universitario de Valencia, Spain; De Roy, Prof., Principal Investigator — Cliniques Universitaires de Mont-Godinne, Yvoir, Belgium; Renato Ricci, Dr., Principal Investigator — San Filippo Neri Hospital, Rome, Italy; Gianluca Botto, Dr., Principal Investigator — Como S. Anna Hospital, Como, Italy; Milan Kozak, Dr., Principal Investigator — Fakultní nemocnice Brno Bohunice, Brno, Czech Republic
Locations (1):
- Medtronic Bakken Research Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Ricci RP, Botto GL, Benezet JM, Nielsen JC, De Roy L, Piot O, Quesada A, Quaglione R, Vaccari D, Mangoni L, Grammatico A, Kozak M; PreFER MVP Investigators. Association between ventricular pacing and persistent atrial fibrillation in patients indicated to elective pacemaker replacement: Results of the Prefer for Elective Replacement MVP (PreFER MVP) randomized study. Heart Rhythm. 2015 Nov;12(11):2239-46. doi: 10.1016/j.hrthm.2015.06.041. Epub 2015 Jun 30. PMID 26142300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start February 2006; last patient enrolled in August 2009.
Pre-assignment Details: Patients were electronically randomized. 25 patients were excluded from analysis due to double entry (7) or no evidence of Patient Informed Consent Form (PIC) signed (18).
Period: Overall Study
Arm/Group | MVP ON | MVP OFF
Started | 299 | 306
Completed | 263 | 265
Not Completed | 36 | 41
Not completed — Lost to Follow-up | 9 | 16
Not completed — Physician Decision | 23 | 17
Not completed — Withdrawal by Subject | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVP ON | MVP OFF | Total
Number analyzed (Participants) | 299 | 306 | 605
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (10.9) | 74.3 (10.8) | 74.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 115 | 240
  Male | 174 | 191 | 365

OUTCOME MEASURES:

1. Primary Outcome: Time to Event Analysis: Number of Patients Who Experienced the First Cardiovascular Hospitalization Within 2 Years Post-implant
Description: Time to first event of cardiovascular (CV) hospitalization from implant to 2 years post-implant.
  Hospitalization is defined as:
  * admission to hospital involving one overnight stay or
  * emergency room / office visits that result in cardioversions or acute treatment of worsened cardiac condition
  Cardiovascular is defined as new or worsening:
  * heart failure (HF),
  * angina,
  * myocardial infarction (MI),
  * any arrhythmia,
  * stroke,
  * transient ischemic attack (TIA),
  * acute peripheral vascular emergencies,
  * pulmonary embolism.
Time Frame: Implant to 2 years post-implant
Population: Patients indicated for Implantable Pulse Generator (IPG) or Implantable Cardioverter Defibrillator (ICD) replacement with a history of right ventricular pacing > 40%, to be allocated to either Managed Ventricular Pacing (MVP) programming, or conventional dual chamber programming (DDD) without MVP
Measure: Number; unit: number of participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
number of participants | 43 | 40
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Analysis:Time to first cardiovascular hospitalization (CV hosp) H0:freedom from CV hosp MVP=freedom from CV hosp DDD (dual chamber conventional pacing) Ha:freedom from CV hosp MVP≠freedom from CV hosp DDD Power calculation: The study is designed to detect a difference event-free survival after 2 years of 5.5 % absolute, going from 91.5% to 97%. Test=two-sided alpha=0.05 power=80% 1:1 randomization n=600; Test type: Superiority or Other; p = 0.72, Log Rank; Hazard Ratio (HR) = 0.927, 95% CI 2-sided [0.612 to 1.405] — Hospitalization:hospital admission with overnight stay;ER/office visits with cardioversions;acute treatment of worsened cardiac condition CV:new/worsening HF,angina,MI,arrhythmia,stroke, TIA,acute peripheral vascular emergencies,pulmonary embolism

2. Secondary Outcome: Time to Event Analysis: Number of Patients Who Experienced Death or First Cardiovascular (CV) Hospitalization Within 2 Years Post-implant.
Description: Time to first event of death or cardiovascular (CV) hospitalization from implant to 2 years post-implant
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
participants
  Death or CV hospitalization at 1 year | 33 | 30
  Death or CV hospitalization at 2 years | 66 | 57
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Analysis:Time to first all cause death or cardiovascular hospitalization H0:freedom from death or CV hospitalization=freedom from death or CV hospitalization Ha:freedom from death or CV hospitalization≠freedom from death or CV hospitalization; Test type: Superiority or Other; p = 0.48, Log Rank; Hazard Ratio (HR) = 1.127, 95% CI 2-sided [0.808 to 1.570]

3. Secondary Outcome: Time to Event Analysis: Number of Patients With Persistent AT/AF Within 2 Years Post-implant
Description: Time to first event of atrial tachycardia/ atrial fibrillation (AT/AF) fulfilling one of the following criteria:
  * 7 days in a row with device diagnostic showing 20 or more hours in AT/AF or
  * a cardioversion was done to terminate AT/AF or
  * the patient is during 2 consecutive follow-up (FU) visits in AT/AF
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
participants
  Persistent AT/AF at 1 year | 27 | 17
  Persistent AT/AF at 2 years | 41 | 30
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Analysis:Time to first persistent AT/AF H0:freedom from persistent AT/AF=freedom from persistent AT/AF Ha:freedom from persistent AT/AF≠freedom from persistent AT/AF; Test type: Superiority or Other; p = 0.08, Log Rank; Hazard Ratio (HR) = 1.521, 95% CI 2-sided [0.954 to 2.424]

4. Secondary Outcome: Time to Event Analysis: Number of Patients With Permanent AF Within 2 Years Post-implant
Description: Time to development of permanent AF fulfilling one of the following criteria:
  * 7 days in a row with device diagnostic showing 20 or more hours in AT/AF and cardioversion failed or
  * 7 days in a row with device diagnostic showing 20 or more hours in AT/AF and the investigator decides not to cardiovert the patient
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
participants
  Permanent AF at 1 year | 8 | 3
  Permanent AF at 2 years | 11 | 8
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Analysis:Time to permanent AF H0:freedom from permanent AF=freedom from permanent AF Ha:freedom from permanent AF≠freedom from permanent AF; Test type: Superiority or Other; p = 0.44, Log Rank; Hazard Ratio (HR) = 1.425, 95% CI 2-sided [0.573 to 3.543]

5. Secondary Outcome: Ventricular Pacing Percentage
Description: Endpoint: Cumulative percentage ventricular pacing documented in the device memory
Time Frame: Implant to 2 years post-implant
Measure: Median (Inter-Quartile Range); unit: Percentage Ventricular Pacing
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
Percentage Ventricular Pacing | 5 [1 to 41] | 86 [40 to 98]
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Analysis:Wilcoxon Test for Comparison of Percentage of Ventricular Pacing (%VP) During Followup by Randomization Arm H0:distribution %VP MVP=distribution %VP DDD Ha:distribution %VP MVP≠distribution %VP DDD Ha:; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF,%) Over 2 Years Time
Description: Endpoint: LVEF (%) difference between 2 year post implant and baseline
Time Frame: Implant to 2 years post-implant
Measure: Mean (Standard Deviation); unit: LVEF (%) difference
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
LVEF (%) difference | -1.2 (10.5) | 1.4 (9.5)
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Test type: Superiority or Other; p = 0.048, Regression, Linear

7. Secondary Outcome: Change in New York Heart Association (NYHA) Functional Class
Description: Endpoint: NYHA classification at Baseline, one year and 2 year post-implant. (Class I is considered a better category and Class IV is considered worse) I Patients with cardiac disease but resulting in no limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea or anginal pain.
  II Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea or anginal pain.
  III Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea or anginal pain.
  IV Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: Baseline, one year and 2 year post-implant
Measure: Number; unit: Participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
Participants
  No Heart Failure (Baseline) | 64 | 92
  Class I (Baseline) | 99 | 87
  Class II (Baseline) | 108 | 108
  Class III (Baseline) | 19 | 9
  Class IV (Baseline) | 1 | 3
  No Heart Failure (12-months) | 67 | 71
  Class I (12-months) | 69 | 72
  Class II (12-months) | 97 | 86
  Class III (12-months) | 5 | 10
  Class IV (12-months) | 0 | 2
  No Heart Failure (24-months) | 53 | 73
  Class I (24-months) | 68 | 69
  Class II (24-months) | 83 | 69
  Class III (24-months) | 11 | 9
  Class IV (24-months) | 0 | 1

8. Secondary Outcome: Change in Use of Anticoagulation
Description: Endpoint: Use of Anticoagulation at enrollment and every follow-up visit
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
participants
  Patients with Medication Records (Baseline) | 298 | 304
  Patients Using Anticoagulants (Baseline) | 75 | 72
  Patients with Medication Records (1-month) | 271 | 285
  Patients Changing Anticoagulants Use (1-month) | 24 | 21
  Patients with Medication Records (12-months) | 246 | 257
  Patients Changing Anticoagulants Use (12-months) | 28 | 31
  Patients with Medication Records (24-months) | 226 | 231
  Patients Changing Anticoagulants Use (24-months) | 27 | 33
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Analysis:Repeated measures logistic regression; Test type: Superiority or Other; p = 0.78, Repeated measures logistic regression

9. Secondary Outcome: Change in the Use of Cardiovascular Medication Over Time
Description: Endpoint: Use of Diuretics, ACE Inhibitors, Beta-Blockers, digitalis, calcium antagonists and antiarrhythmic drugs at enrollment, and 1month, 12 months, and 24 mnths after implant
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 298 | 304
participants
  Beta-blockers (Baseline), n=298, 304 | 129 | 116
  Digitalis/digoxin (Baseline), n=298, 304 | 26 | 30
  Calcium antagonists (Baseline), n=298, 304 | 54 | 63
  Antiarrhythmic drugs (Baseline), n=298, 304 | 81 | 103
  Beta-blockers (1-month), n=271, 285 | 117 | 111
  Digitalis/digoxin (1-month), n=271, 285 | 24 | 28
  Calcium antagonists (1-month), n=271, 285 | 49 | 60
  Antiarrhythmic drugs (1-month), n=271, 285 | 75 | 98
  Beta-blockers (12-months), n=246, 257 | 108 | 105
  Digitalis/digoxin (12-months), n=246, 257 | 22 | 26
  Calcium antagonists (12-months), n=246, 257 | 46 | 52
  Antiarrhythmic drugs (12-months), n=246, 257 | 67 | 88
  Beta-blockers (24-months), n=226, 231 | 104 | 93
  Digitalis/digoxin (24-months), n=226, 231 | 20 | 22
  Calcium antagonists (24-months), n=226, 231 | 36 | 47
  Antiarrhythmic drugs (24-month), n=226, 231 | 58 | 76
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Analysis:Repeated measures logistic regression H0:Change in Beta-blockers=Change in Beta-blockers Ha:Change in Beta-blockers≠Change in Beta-blockers; Test type: Superiority or Other; p = 0.34, Regression, Logistic
Statistical Analysis 2: Comparison: MVP ON vs MVP OFF; Analysis:Repeated measures logistic regression H0:Change in Digitalis/digoxin=Change in Digitalis/digoxin Ha:Change in Digitalis/digoxin≠Change in Digitalis/digoxin; Test type: Superiority or Other; p = 0.65, Regression, Logistic
Statistical Analysis 3: Comparison: MVP ON vs MVP OFF; Analysis:Repeated measures logistic regression H0:Change in Calcium antagonists=Change in Calcium antagonists Ha:Change in Calcium antagonists≠Change in Calcium antagonists; Test type: Superiority or Other; p = 0.55, Regression, Logistic
Statistical Analysis 4: Comparison: MVP ON vs MVP OFF; Analysis:Repeated measures logistic regression H0:Change in Antiarrhythmic drug=Change in Antiarrhythmic drug Ha:Change in Antiarrhythmic drug≠Change in Antiarrhythmic drug; Test type: Superiority or Other; p = 0.53, Regression, Logistic

10. Secondary Outcome: Incidence of High Voltage Therapies
Description: Endpoint: A high voltage therapy delivered
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
participants | 1 | 3

11. Secondary Outcome: Time to Event Analysis: Number of Patients Who Died Within 2 Years Post-implant
Description: Time to patient death from any cause
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP Off
Number analyzed (Participants) | 299 | 306
participants
  All-Cause Death at 1 year | 17 | 7
  All-Cause Death at 2 years | 31 | 22
Statistical Analysis 1: Comparison: MVP ON vs MVP Off; Analysis:Time to all-cause death H0:survival MVP ON=survival MVP OFF Ha:survival MVP ON≠survival MVP OFF; Test type: Superiority or Other; p = 0.33, Log Rank; Hazard Ratio (HR) = 1.243, 95% CI 2-sided [0.803 to 1.923]

12. Secondary Outcome: Stroke
Description: Endpoint: Stroke
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
participants
  Stroke at 1 year | 3 | 4
  Stroke at 2 years | 4 | 6
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Test type: Superiority or Other; p = 0.24, Log Rank; Hazard Ratio (HR) = 0.492, 95% CI 2-sided [0.148 to 1.637]

13. Secondary Outcome: Number of Cardiovascular Related Hospitalizations
Description: Endpoint: Number of Cardiovascular hospitalizations per subject
Time Frame: Implant to 4 years post-implant
Population: All participants were followed for 4 years. Those not hospitalized were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: Number of CV Hospitalizations
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 53 | 46
Number of CV Hospitalizations | 1.0 [1 to 2] | 1.0 [1 to 2]
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Statistical test for Number of subjects with CV hospitalization; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Duration of Cardiovascular Related Hospitalizations
Description: Endpoint: Duration of Cardiovascular Hospitalizations per subject
Time Frame: Implant to 4 years post-implant
Population: All participants were followed for 4 years. Those not hospitalized were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: Days of CV hospitalizations
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 53 | 46
Days of CV hospitalizations | 7.0 [4 to 12] | 7.5 [3 to 14]

15. Secondary Outcome: Incidence of Class I Pacemaker (Implantable Pulse Generator = IPG) Indication in Implantable Cardioverter Defibrillator (ICD) Patients
Description: Endpoint: Patient implanted with a replacement ICD developing a class 1 pacemaker indication
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 28 | 21
participants | 0 | 0

16. Secondary Outcome: Change in PR Interval, Change in QRS Duration and Change in P-wave Duration
Description: Endpoint: Change in PR interval, Change in QRS duration and Change in P-wave duration evaluated at enrollment and 24 Month FU
Time Frame: Implant to 2 years post-implant
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
milliseconds
  PR interval (ms) difference 24 month-baseline | 11.6 (60.9) | 10.8 (63.6)
  QRS duration (ms) difference: 24 month-baseline | 2.6 (32.4) | 10.8 (41.8)
  P-wave duration (ms) difference: 24 month-baseline | 5.2 (41.2) | 1.1 (38.4)
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; H0:Change in P-R interval=Change in P-R interval Ha:Change in P-R interval≠Change in P-R interval; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: MVP ON vs MVP OFF; H0:Change in QRS duration=Change in QRS duration Ha:Change in QRS duration≠Change in QRS duration; Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: MVP ON vs MVP OFF; H0:Change in P-wave duration=Change in P-wave duration Ha:Change in P-wave duration≠Change in P-wave duration; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Patient Symptoms
Description: Endpoint: Symptoms evaluated at enrollment, 12 months and 24 months followup
Time Frame: Implant to 2 years post-implant
Measure: Number; unit: participants
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 299 | 306
participants
  No symptoms (baseline) | 175 | 193
  Chest pain (baseline) | 24 | 15
  Dyspnea (baseline) | 65 | 59
  Dizziness/presyncope (baseline) | 32 | 27
  No Symptoms (12 months) | 175 | 184
  Chest pain (12 months) | 11 | 12
  Dyspnea (12 months) | 36 | 38
  Dizziness/presyncope (12 months) | 9 | 17
  No Symptoms (24 months) | 158 | 160
  Chest pain (24 months | 15 | 10
  Dyspnea (24 months) | 39 | 40
  Dizziness/presyncope (24 months) | 8 | 15
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; No Symptoms (Baseline); Test type: Superiority or Other; p = 0.24, Fisher Exact
Statistical Analysis 2: Comparison: MVP ON vs MVP OFF; No Symptoms (12 months); Test type: Superiority or Other; p = 0.92, Fisher Exact
Statistical Analysis 3: Comparison: MVP ON vs MVP OFF; No Symptoms (24 Months); Test type: Superiority or Other; p = 1.0, Fisher Exact

18. Secondary Outcome: Atrial Pacing Percentage
Description: Endpoint: Cumulative percentage atrial pacing documented in the device memory
Time Frame: 2 years post-implant
Measure: Median (Inter-Quartile Range); unit: percentage atrial pacing
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 279 | 283
percentage atrial pacing | 68 [36 to 94] | 78 [47 to 95]
Statistical Analysis 1: Comparison: MVP ON vs MVP OFF; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Health State
Description: Endpoint: Health State evaluation with the EQ-5D questionnaire (range 0-100) . A measure of 100 is better and a measure of 0 is worse.
Time Frame: 2 years post-implant
Population: Patients with health evaluation completed at 24 months follow-up
Measure: Mean (Standard Deviation); unit: units on a Health State scale
Arm/Group | MVP ON | MVP OFF
Number analyzed (Participants) | 219 | 224
units on a Health State scale | 70.6 (17.2) | 70.3 (16.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until study closure. The following abbreviations are used in the additional description: SAE: serious adverse event. (S)ADE: (serious) adverse device effect. PE: primary endpoint.
Description: The following adverse events had to be reported:
  * SAEs (for study purposes also included: 1) cardioversion and 2) emergency room / office visits resulting in acute treatment for worsened cardiac condition
  * Deaths
  * (S)ADE
  The PE committee adjudicated all reported AEs per the primary objective. No further classification has been done.
Arm/Group | MVP ON | MVP OFF
Serious Adverse Events (participants affected / at risk) | 85/299 | 72/306
Other Adverse Events (participants affected / at risk) | 32/299 | 31/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVP ON (N=299) | MVP OFF (N=306)
First cardiovascular hospitalization within 2 years after implant (Cardiac disorders) | 43 (43) | 40 (40) — Hospitalization (including emergency room) for cardiovascular causes: new or worsening heart failure, angina, myocardial infarction, any arrhythmia, stroke, transient ischemic attack, acute peripheral vascular emergencies, pulmonary embolism.
Cardioversion within 2 years after implant (Cardiac disorders) | 11 (15) | 9 (13) — Cardioversion medically or electrically
Stroke within 2 years after implant (Nervous system disorders) | 4 (4) | 6 (6) — Stroke
Death from any cause within 2 years after implant (General disorders) | 31 (31) | 22 (22) — All cause death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVP ON (N=299) | MVP OFF (N=306)
Non serious adverse events up to 2 years follow-up (General disorders) | 32 (47) | 31 (39) — All reported adverse events which were not serious

LIMITATIONS AND CAVEATS:
Atrial pacing % was not collected at implant, device programming in the MVP off arm was more often non-compliant than in MVP on arm, and 25% of the case report forms were sent without device data, possibly influencing device data related objectives

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days